CLINICAL TRIAL: NCT00339976
Title: Ascertainment of Death in ALS Patients
Brief Title: Exposure to Neurotoxins as Risk Factors for Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902275; 02-E-N275
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-04-21

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: Case-Control Study; Death Certificates; National Death Index; Cause of Death Information; Lead Exposure; Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

SUMMARY:
This study is a follow-up to an earlier study that examined the relationship of This study will examine whether exposure to neurotoxins, such as lead, mercury, solvents, and pesticides, can contribute to amyotrophic lateral sclerosis (ALS), also known as Lou Gehrig's disease. The cause of this degenerative disease of the brain and spinal cord is not well understood. Some studies suggest that exposure to environmental neurotoxins may increase its risk. This follow-up study will examine the relationship of neurotoxin exposure to the interval between the diagnosis of ALS and death. It will also examine the possible roles of genetics, lifestyle and dietary factors in the disease. Information on ALS patients previously enrolled in the study will be used to examine this relationship. No new individuals will be enrolled in the study.

DETAILED DESCRIPTION:
Objective: The objective of this proposal is linkage with the National Death Index (NDI) for cases from a study that was conducted in the early 1990's. The purpose of the initial study was to examine the role that lead and other exposures, including mercury and solvents, play in the etiology of amyotrophic lateral sclerosis (ALS).

Study population: The study involved 110 ALS cases and 256 population based controls, recruited in New England between 1993 and 1996. Data collection involved an interview, blood collection, and measurement of bone lead using x-ray fluorescence.

Design and outcome parameters: The results of this study suggested that lead exposure was a risk factor for ALS. Compared to controls, cases were more likely to have occupational lead exposure, and both blood and bone lead levels were higher in cases. We are presently analyzing data on other neurotoxic exposures including mercury, solvents, and pesticides. In order to investigate prognosis, we would like to determine the date of death by searching the National Death Index. This information will enable us to evaluate the relationship of neurotoxic exposures to ALS prognosis.

ELIGIBILITY:
* INCLUSION CRITERIA:

The purpose of the NDI search will be to verify death and obtain date and cause of death information for the study participants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 2002-08-06; Study Completion 2008-04-21

CONTACTS AND LOCATIONS:
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Bharucha NE, Schoenberg BS, Raven RH, Pickle LW, Byar DP, Mason TJ. Geographic distribution of motor neuron disease and correlation with possible etiologic factors. Neurology. 1983 Jul;33(7):911-5. doi: 10.1212/wnl.33.7.911. PMID 6683374